CLINICAL TRIAL: NCT01901289
Title: Zilver® PTX® Drug-Eluting Peripheral Stent Post-Approval Study
Brief Title: Zilver® PTX® V Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-004
Record Dates: First submitted 2013-07-08; First posted 2013-07-17 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Vascular Disease; Femoral Artery; Popliteal Artery; Drug-Eluting Stent
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No

ARMS (1):
- Drug-Eluting Stent (Experimental)
  Interventions: Device: Zilver® PTX® Drug-Eluting Peripheral Stent

INTERVENTIONS:
Device: Zilver® PTX® Drug-Eluting Peripheral Stent — Treatment of symptomatic vascular disease of the native above-the-knee femoropopliteal arteries.

SUMMARY:
The Zilver® PTX® V Clinical Study is a post-market clinical trial required by the US FDA to provide continued evaluation of the safety and effectiveness of the Zilver PTX Drug-Eluting Peripheral Stent in treatment of narrowing of the femoropopliteal arteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient has signed and dated the informed consent.
* Patient has symptomatic vascular disease of the native above-the-knee femoropopliteal arteries.
* Patient agrees to return for the required follow-up assessments.

Exclusion Criteria:

* Patient is < 18 years of age.
* Patient has significant stenosis of inflow tract not successfully treated before this procedure.
* Patient lacks at least one patent vessel of runoff with < 50% stenosis throughout its course.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-08; Primary Completion 2016-11-18 (Actual); Study Completion 2021-02-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - VA Palo Alto Health Care System, Palo Alto, California
  - Stanford University Medical School, Stanford, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Bayview Medical Center, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - New York-Presbyterian/ Weill Cornell Medical Center, New York, New York
  - OhioHealth Research Institute, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - Holy Spirit Hospital, Camp Hill, Pennsylvania
  - South Carolina Heart Center, Columbia, South Carolina
  - Greenville Hospital System, Greenville, South Carolina
  - Holston Valley Hospital, Kingsport, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after final report has been distributed and ending 5 years after final report has been distributed. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.

REFERENCES:
- [Derived] Dake MD, Fanelli F, Lottes AE, O'Leary EE, Reichert H, Jiang X, Fu W, Iida O, Zen K, Schermerhorn M, Zeller T, Ansel GM. Prediction Model for Freedom from TLR from a Multi-study Analysis of Long-Term Results with the Zilver PTX Drug-Eluting Peripheral Stent. Cardiovasc Intervent Radiol. 2021 Feb;44(2):196-206. doi: 10.1007/s00270-020-02648-6. Epub 2020 Oct 6. PMID 33025243

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug-Eluting Stent
Started | 200
12-Month Follow-up | 194
Completed | 115
Not Completed | 85
Not completed — Death | 32
Not completed — Lost to Follow-up | 16
Not completed — Withdrawal by Subject | 35
Not completed — Other type of endpoint met | 2

BASELINE CHARACTERISTICS:
Arm/Group | Drug-Eluting Stent
Number analyzed (Participants) | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2
  Black | 22
  Black/Caucasian or White | 1
  Caucasian or White | 165
  Hispanic or Latino | 10
Region of Enrollment [Number; unit: participants]
  United States | 200
Diabetes [Count of Participants; unit: Participants] | 92
Smoking Status [Count of Participants; unit: Participants]
  Never smoked | 31
  Quit smoking | 86
  Still smoking | 83
Hypercholesterolemia [Count of Participants; unit: Participants] | 173

OUTCOME MEASURES:

1. Primary Outcome: Patients Without Target Lesion Revascularization (TLR)
Description: A reintervention performed for ≥ 50 % diameter stenosis within ± 5 mm proximal and /or distal to the target lesion after documentation of recurrent clinical symptoms of peripheral arterial disease (PAD) following the initial procedure.
Time Frame: 1 year
Population: The result was calculated using the Kaplan-Meier method (with Greenwood's formula for standard error).
Measure: Count of Participants; unit: Participants
Arm/Group | Drug-Eluting Stent
Number analyzed (Participants) | 200
Participants | 186
Statistical Analysis 1: Comparison: Drug-Eluting Stent; Test type: Other; Cumulative Probability = 0.927, 95% CI 2-sided [0.881 to 0.956], Standard Error of Mean 0.019 — The estimate of the variance of the Kaplan-Meier estimate used the methods described by Peto et al

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Drug-Eluting Stent
All-Cause Mortality (participants affected / at risk) | 32/200
Serious Adverse Events (participants affected / at risk) | 154/200
Other Adverse Events (participants affected / at risk) | 46/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-Eluting Stent (N=200)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Bandaemia (Blood and lymphatic system disorders) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 4 (4)
Angina unstable (Cardiac disorders) | 4 (4)
Arrhythmia (Cardiac disorders) | 7 (7)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrial flutter (Cardiac disorders) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 2 (3)
Cardiac failure (Cardiac disorders) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 16 (25)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 5 (5)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 11 (13)
Myocardial ischaemia (Cardiac disorders) | 20 (26)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Femoral hernia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 13 (16)
Ileus (Gastrointestinal disorders) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 3 (4)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Mesenteric arterial occlusion (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2)
Rectal prolapse (Gastrointestinal disorders) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Volvulus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 7 (12)
Fatigue (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (6)
Pain (General disorders) | 1 (1)
Physical deconditioning (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Stent-graft endoleak (General disorders) | 1 (1)
Vascular stent stenosis (General disorders) | 4 (4)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Gallbladder polyp (Hepatobiliary disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic mass (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 2 (2)
Bacterial colitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 6 (6)
Cellulitis streptococcal (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 2 (2)
Device related sepsis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Emphysematous cholecystitis (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Endocarditis (Infections and infestations) | 2 (2)
Endocarditis bacterial (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 5 (8)
Gastroenteritis (Infections and infestations) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Intervertebral discitis (Infections and infestations) | 1 (1)
Large intestine infection (Infections and infestations) | 1 (1)
Meningitis bacterial (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 2 (2)
Parotitis (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (3)
Pneumonia (Infections and infestations) | 19 (25)
Postoperative wound infection (Infections and infestations) | 2 (2)
Pseudomonal bacteraemia (Infections and infestations) | 1 (3)
Pyelonephritis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 5 (5)
Sinusitis (Infections and infestations) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3)
Streptococcal bacteraemia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 10 (12)
Vascular access site infection (Infections and infestations) | 1 (1)
West Nile viral infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 2 (3)
Arterial bypass stenosis (Injury, poisoning and procedural complications) | 1 (1)
Arterial bypass thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Arterial restenosis (Injury, poisoning and procedural complications) | 3 (3)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (2)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2 (2)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 (1)
Carotid artery restenosis (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 8 (11)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 39 (60)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Restenosis (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (3)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (1)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Catheterisation cardiac abnormal (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Troponin (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (4)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung adenocarcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant respiratory tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Rectosigmoid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 4 (6)
Cerebrovascular accident (Nervous system disorders) | 9 (9)
Dizziness (Nervous system disorders) | 3 (3)
Encephalopathy (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 6 (6)
Toxic encephalopathy (Nervous system disorders) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Device damage (Product Issues) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 3 (3)
Substance abuse (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (9)
Bladder mass (Renal and urinary disorders) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 10 (12)
Urinary retention (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1)
Penis disorder (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 8 (16)
Debridement (Surgical and medical procedures) | 1 (1)
Dialysis device insertion (Surgical and medical procedures) | 1 (1)
Medical device battery replacement (Surgical and medical procedures) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1)
Mitral valve repair (Surgical and medical procedures) | 1 (1)
Rotator cuff repair (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 3 (3)
Aortic stenosis (Vascular disorders) | 2 (2)
Arterial stenosis (Vascular disorders) | 1 (1)
Atheroembolism (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Hypertensive emergency (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Hypovolaemic shock (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 32 (48)
Ischaemia (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral artery dissection (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 17 (22)
Peripheral artery stenosis (Vascular disorders) | 4 (4)
Peripheral artery thrombosis (Vascular disorders) | 10 (19)
Peripheral coldness (Vascular disorders) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 2 (3)
Peripheral vascular disorder (Vascular disorders) | 2 (3)
Steal syndrome (Vascular disorders) | 2 (2)
Subclavian artery stenosis (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug-Eluting Stent (N=200)
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 16 (16)
Intermittent claudication (Vascular disorders) | 32 (45)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications from PI prior to public release and can embargo communications of trial results between 60 and 180 days from the time submitted to the sponsor for review. The sponsor can embargo publications until the sponsor has published results or 180 days has elapsed after study closure at all participating sites. The sponsor cannot restrict publication but can require changes to protect sponsor's intellectual property rights or other confidential information.